CLINICAL TRIAL: NCT03100474
Title: Global Registry: ExAblate 4000 Transcranial MR Guided Focused Ultrasound (TcMRgFUS) of Neurological Disorders:
Brief Title: Global Registry: ExAblate Neuro MR Guided Focused Ultrasound (MRgFUS) of Neurological Disorders:
Status: Active, not recruiting | Type: Observational
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: ND001
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor; Parkinson's Disease; Movement Disorders; Neuropathic Pain
Keywords: tremor; Parkinson's; movement; neuropathic; pain
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Movement Disorders; Neuralgia; Tremor; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A global post approval study to collect safety and effectiveness data related to ExAblate Neuro for the treatment of certain disorders such as Essential Tremor, Parkinson's Movement Disorders, or Neuropathic Pain within the thalamus and/or pallidum.

DETAILED DESCRIPTION:
A global, multi-center, open-label, observational registry to capture safety and effectiveness data related to ExAblate Neuro, an MRI guided focused ultrasound device designed to lesion tissue deep within the brain using sound waves without the need for craniotomy. This registry includes certain regional and country specific approved thalamotomy and pallidotomy procedures using ExAblate Neuro for the treatment of various neurologic disorders such as essential tremor, Parkinson's movement disorders, and neuropathic pain. Treatment targets/indications are country/region dependent based on approved labeling within that region.

ELIGIBILITY:
Inclusion Criteria:

* Meets labeling indication for use per information for prescribers
* Target is accessible by Focused Ultrasound per treatment planning parameters

Exclusion Criteria:

* Do not agree to participate or who are unlikely to participate over an extended period of time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients suffering from clinically diagnosed neurologic disorders that can be
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor | 5 year
  CRST

CONTACTS AND LOCATIONS:
Overall Officials: Howard Eisenberg, MD, Principal Investigator — University of Maryland
Locations (9):
- United States (5):
  - Stanford University, Stanford, California
  - University of Maryland, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
- Sunnybrook, Toronto, Ontario, Canada
- Israel (2):
  - Rambam Healthcare Campus, Haifa
  - Sheba Medical Center, Ramat Gan
- Chang Bing Show Chwan Memorial Hospital, Chang-hua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared via request from the publication committee. Active site participants will have access; however, it has not been decided when or if data will be shared with researchers not participating on this registry.